CLINICAL TRIAL: NCT03426761
Title: Dalbavancin For The Treatment Of Gram Positive Osteomyelitis Or Joint Infections Including Prosthetic Hip Or Knee Infections
Brief Title: Dalbavancin For The Treatment of Gram Positive Osteoarticular Infections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Infectious Diseases Physicians, Inc. (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2017-10117
Record Dates: First submitted 2018-01-26; First posted 2018-02-08 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Bone Infection; Osteomyelitis; Septic Arthritis; Joint Infection; Prosthetic Joint Infection
MeSH Terms: conditions — Osteomyelitis; Arthritis, Infectious | interventions — dalbavancin; Vancomycin; Daptomycin; Nafcillin; Cefazolin

STUDY DESIGN:
Intervention Model Description: Since it's a pilot study, the sample size is fixed (n = 50). The sample size were not selected based on statistical criteria. However, we would need to know what would be the detectable effect size.
  ∆^2=((z_(α/2)+z_β )^2 (σ_1^2+σ_2^2 ))/n
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dalbavancin (Experimental): Dalbavancin 1,500mg intravenously every fourteen days for two to four infusions
  Interventions: Drug: Dalbavancin
- Standard of Care (Active Comparator): Standard of care intravenous antibiotic based on microbiology susceptibility testing. Infusions may be one to three times daily for three to eight weeks. Examples of standard of care include vancomycin, daptomycin, nafcillin, cefazolin.
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Dalbavancin — Dalbavancin 1,500mg intravenously every fourteen days for two to four infusions
  Other Names: Dalvance; Xydalba; Zevan
  Arms: Dalbavancin
Drug: Vancomycin — Examples of standard of care arm; infusions one to three times per day depending on the antibiotic for a total of three to eight weeks
  Other Names: Daptomycin; Nafcillin; Cefazolin
  Arms: Standard of Care

SUMMARY:
Because of its prolonged terminal half-life, dalbavancin is an extremely attractive option in treating Gram-positive infections caused by S. aureus including MRSA, and streptococcal species. Systemic bacterial infections due to Staphylococci such as osteomyelitis and septic arthritis, are conditions which require prolonged IV therapy, typically for at least 3-6 weeks, though sometimes more. Due to dalbavancin's prolonged terminal half-life, it may offer the opportunity to substantially reduce costs and morbidity in native joint and prosthetic joint infections with one infusion every fourteen days until completion of therapy.

DETAILED DESCRIPTION:
Dalbavancin, currently FDA approved for the treatment of skin and soft tissue infections (SSTI), is a lipoglycopedptide with bactericidal activity in vitro against Staphylococcus aureus, including MRSA and VISA strains, and Streptococcus pyogenes. Its bactericidal action results primarily from inhibition of cell-wall biosynthesis, specifically the prevention of N-acetylmuramic acid (NAM) and N-acetylglucosamine (NAG)-peptide subunits incorporation into the peptidoglycan matrix. Dalbavancin alters bacterial-cell-membrane permeability and RNA synthesis. It is highly protein bound, primarily to albumin, with a half-life of 346 hours. Approximately 33% of unchanged drug is excreted in the urine, 20% via feces and 12% as the minor metabolite, hydroxyl-dalbavancin. There is minimal potential for drug-drug interactions; it is not a substrate, inducer or inhibitor of hepatic CYP450 isoenzymes and the administration of CYP450 substrates, inhibitors or inducers does not affect its clearance rate. In SSTI trials, Dalbavancin was demonstrated to be non-inferior to vancomycin and linezolid.

Prosthetic joint infections (PJI) are an emerging health problem. Although the incidence of these infections is historically low (approximately 0.5%-1.0of implants), because of the rapid increase in the number of hip, knee and other joint implants, the absolute number of cases of infection is increasing. In 2010, 332,000 hip joints and 719,000 knee joints were implanted. This alone conservatively translates to 5,000-10,000 cases, with an economic impact of $1 billion. Management of PJI is particularly challenging because long term antibiotic therapy in most cases is accompanied by removal of the prosthesis and re-implantation.

For long term antimicrobial administration, current standard of care requires a peripherally inserted central catheter (PICC) or other indwelling intravascular catheter, and daily/multiple daily infusions. There is substantial cost of maintaining the intravascular access, drugs, home health care and monitoring, as well as the infection risk of the chronic indwelling line which is being accessed frequently. There is a clear need for alternative care models to the current approach. Dalbavancin, because of its activity profile against Gram-positive organisms and its pharmacokinetics which would allow weekly or every other week dosing, is a favorable option. This option would eliminate the need for long term IV access, because at most, weekly IV infusions would be performed.

In terms of bone infection, dalbavancin has favorable pharmacokinetic properties. A PK study performed in subjects undergoing elective orthopedic surgery found that dalbavancin (dosed at 1000mg IV at enrollment and then 500mg weekly for up to 7 weeks) maintained levels in cortical bone at bactericidal levels , at >50X the MIC of typical staphylococcal organism (including MRSA). Animal studies in a rat osteomyelitis model also found that dalvabancin was comparable to vancomycin. Because of these same PK properties, dalbavancin offers the opportunity to substantially reduce costs and morbidity in native joint and prosthetic joint infections.

This is a two-center, randomized, open label trial of dalbavancin versus standard intravenous therapy control comparator in the treatment of subjects with gram positive native joint or prosthetic joint infections. The primary outcome variable is clinical cure at day 42 after start of treatment in all randomized patients. Safety and tolerability will also be assessed throughout the study period via laboratory measurements and AE monitoring. Additionally, clinical response will be measured by patient reported outcomes with change from baseline symptoms and by Quality of Life questionnaire.

Eligible subjects with confirmed gram positive joint infections, will be randomized in a ratio of 2:1 to receive open label dalbavancin or standard IV therapy. Standard IV therapy will depend on the antibiotic susceptibility of the causative pathogen. Subjects randomized to dalbavancin may have received standard of care therapy for no more than 120 hours prior to first dalbavancin dose. Subjects randomized to standard of care can continue with treatment course if already started, or receive the first dose at the baseline visit.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained from the patient (if possible) or from either the caregiver or legally authorized representative (if different from the caregiver) before the initiation of any study specific procedures.
2. Male or female patients, aged 18-80, with the following osteoarticular infections:

   1. Infected shoulder, knee or hip (1st or 2nd episode) as defined by a diagnostic culture positive arthrocentesis
   2. An infected prosthetic shoulder, knee or hip as defined by a diagnostic culture positive arthrocentesis, or intraoperative diagnosis of infection with positive culture; an infected prosthetic knee or hip (1st or 2nd episode). Preoperative diagnosis by diagnostic, culture positive arthrocentesis
3. Demonstrated by a positive culture for one of the following gram positive organisms: Methicillin susceptible Staphyloccocus aureus, methicillin resistant Staphylococcus aureus, Streptococcus pyogenes, Group B streptococcus, Streptococcus anginosus group, Vancomycin susceptible Enterococcus faecalis
4. If female, meet the following criteria:

   1. Not breastfeeding
   2. Not planning to become pregnant during the study
   3. Be surgically sterile, or at least 2-years postmenopausal, or have a negative pregnancy test at Baseline (Visit 1)
   4. If of childbearing potential, agree to be strictly abstinent, or practice 2 of the following effective methods of birth control throughout the study: systemic contraception (e.g., oral contraceptives of estrogen and progestin combinations); depot injection (e.g., Depo-Provera); contraceptive implant (e.g., Norplant, Implanon); transdermally delivered contraceptive (e.g., Ortho Evra); intrauterine device; vaginal contraceptive ring (e.g.,NuvaRing); diaphragm plus spermicide; cervical cap; or male condom plus spermicide; partner vasectomy at least 6 months prior to baseline
5. Vision and hearing (hearing aid permissible) sufficient for compliance with testing procedures

Exclusion Criteria:

1. Subjects with culture proven gram negative infection
2. Concurrent diseases that, in the Investigator's medical judgment, would interfere with the conduct of the study, confound the interpretation of the study results, or endanger the patient's well-being
3. Any other conditions that, in the investigator's opinion, might indicate that the patient is unsuitable for the study, the exception is, if there is a history of such disease but the condition has been stable for at least more than 3 year(s) and the investigator determines that it would not interfere with the patient's participation in the study
4. Current malignancy under treatment with chemotherapeutic agents
5. Any unapproved concomitant medication excluded in section 6.3 that could not be discontinued or switched to an allowable alternative medication before the Baseline (Visit 2)
6. Currently participating in or previously participated in an investigational study of Dalbavancin or treatment with an investigational product within 3 months or 5 half-lives, whichever is longer, of Screening (Visit 1)
7. HIV infection with a CD4 count <200
8. Solid organ transplantation or bone marrow transplantation within 6 months
9. History of severe neutropenia, defined as an absolute neutrophil count (ANC) <500 cells per microliter, in the last three months
10. History of severe liver disease, i.e. Child-Pugh Class C or aspartate aminotransferase (AST) or alanine aminotransferase (ALT) more than five times the upper limit of normal (ULN), in the last three months
11. Positive blood culture in the past 14 days, evidence of multiple sites of joint infection, or evidence of concomitant infections at other body sites related to bacteremia
12. Positive test on a urine drug screening for drugs of abuse, for which the patient does not have prescription
13. History of drug or alcohol abuse that, in the Investigator's medical judgment, would interfere with the conduct of the study
14. History of hypersensitivity reaction to Dalbavancin or other drugs of the same class

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Clinical response (non-failure) to assigned treatment at day #42 | Evaluated at Day 42
  This is defined as the absence of wound drainage, sinus tract formation, fever or joint instability at study day 42, without having switched or extended treatment for any reason. This will be reported as the % of participants from each treatment arm, who are determined to be a treatment responder.

SECONDARY OUTCOMES:
Sustained Clinical Response at day #90 | Evaluated at Day 90
  This is defined as the absence of drainage, sinus tract formation, fever, cellulitis, infectious effusion (culture +) or joint instability.
Sustained Clinical Response at day #180 | Evaluated at Day 180
  This is defined as the absence of drainage, cellulitis, infectious effusion (culture +) or joint instability.
Sustained Clinical Response at day #365 | Evaluated at Day 365
  This is defined as the absence of drainage, cellulitis, infectious effusion (culture +) or joint instability.
CRP Improvement at day #90 | Evaluated at Day 90
  Normalized or, at least 75% reduction from baseline
CRP Improvement at day #180 | Evaluated at Day 180
  Normalized or, at least 75% reduction from baseline
CRP Improvement at day #365 | Evaluated at Day 365
  Normalized or, at least 75% reduction from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Donald Poretz, MD, Principal Investigator — Infectious Diseases Physicians, Inc.
Locations (1):
- Infectious Diseases Physicians, Inc., Annandale, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided
Upon conclusion of the statistical analysis, the study team may write their findings for an infectious disease journal article

REFERENCES:
- See also: Infectious Diseases Physicians, Inc. — http://idphysicians.net